CLINICAL TRIAL: NCT03436056
Title: PembRolIzuMab and Stereotactic Body Radiotherapy In Metastatic Non-small-cell lunG Cancer Patients
Acronym: PRIMING
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: funding pulled
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 4590; NCT03368222 (obsolete NCT alias)
Record Dates: First submitted 2018-01-16; First posted 2018-02-19 (Actual); Results first posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Metastatic Non-small-cell lunG Cancer
Keywords: Non-small-cell lunG cancer; NSCLC; metastatic; pembrolizumab; radiotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasm Metastasis | interventions — Radiosurgery; pembrolizumab

STUDY DESIGN:
Intervention Model Description: Dose Escalation phase with 2 dose levels followed by an Expansion phase
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Dose escalation cohort - DOSE LEVEL 1 (Other): Intervention: One dose pembrolizumab 200 mg (week 1) followed by lung Stereotactic Body Radiotherapy (SBRT) 30 Gy 3 fractions (#) in week 3. Treatment with pembrolizumab 200 mg will be continued given every 3 weeks.
  Interventions: Radiation: Stereotactic Body Radiotherapy (SBRT) 30 Gy 3 fractions (#); Drug: Pembrolizumab
- Dose escalation cohort - DOSE LEVEL 2 (Other): Intervention: One dose of pembrolizumab 200 mg (week 1) followed by lung Stereotactic Body Radiotherapy (SBRT) 54 Gy 3 fractions (#) in week 3. Treatment with pembrolizumab 200 mg will be continued given every 3 weeks.
  Interventions: Radiation: Stereotactic Body Radiotherapy (SBRT) 54 Gy 3 fractions (#); Drug: Pembrolizumab
- Part B - Expansion cohort (Other): Intervention: One dose of pembrolizumab 200 mg (week 1) followed in by lung Stereotactic Body Radiotherapy (SBRT) dosed at the maximum tolerated dose determined in Part A in week 3, dosed at the maximum tolerated dose determined in Part A. Treatment with pembrolizumab 200 mg will be continued given every 3 weeks.
  Interventions: Radiation: Stereotactic Body Radiotherapy (SBRT) dosed at the maximum tolerated dose; Drug: Pembrolizumab

INTERVENTIONS:
Radiation: Stereotactic Body Radiotherapy (SBRT) 30 Gy 3 fractions (#) — Stereotactic Body Radiotherapy (SBRT) dosed at 30 Gy in 3 fractions (#) in week 3
  Arms: Dose escalation cohort - DOSE LEVEL 1
Radiation: Stereotactic Body Radiotherapy (SBRT) 54 Gy 3 fractions (#) — Stereotactic Body Radiotherapy (SBRT) dosed at 54 Gy in 3 fractions (#) in week 3
  Arms: Dose escalation cohort - DOSE LEVEL 2
Radiation: Stereotactic Body Radiotherapy (SBRT) dosed at the maximum tolerated dose — Stereotactic Body Radiotherapy (SBRT) dosed at the maximum tolerated dose (MTD) determined in Part A in week 3
  Arms: Part B - Expansion cohort
Drug: Pembrolizumab — Pembrolizumab in week 1 dosed at 200 mg (prior to SBRT) and then treatment with pembrolizumab will be continued dosed at 200 mg given every 3 weeks.
  Other Names: Keytruda

SUMMARY:
This is a single centre non-randomised open label phase 1 trial of lung SBRT to part of a lung lesion in patients with advanced NSCLC in combination with pembrolizumab. This study will recruit up to 24 patients whose lung cancer has progressed beyond one line of palliative chemotherapy, and an EGFR or ALK inhibitor if an EGFR driver mutation or ALK gene rearrangement is present, respectively, and now requires further palliative systemic treatment.

DETAILED DESCRIPTION:
The study will be conducted in two parts; an initial lung SBRT dose escalation phase (Part A), followed by a lung SBRT dose expansion cohort (Part B). The dose escalation phase is based on a 3+3 design such that patients will be treated in cohorts of 3-6 patients. A maximum of 12 patients will be allocated to one of two doses of lung SBRT in combination with pembrolizumab to determine the MTD, DLTs and RP2D. If there is more than one DLT in cohort 1, this treatment combination will be deemed as being unacceptable, and it would lead to termination of the study. Note, there is no de-escalation in cohort 1. During the dose expansion cohort, 12 patients will have lung SBRT dosed at the RP2D determined during the dose escalation phase in combination with pembrolizumab to obtain additional safety and response data. Maintenance pembrolizumab will continue until disease progression, unacceptable toxicities, the patient withdraws consent to the trial, or the patient has completed 24 months of treatment. A maximum of 24 patients will be treated in the study.

All patients will receive pembrolizumab on cycle (C) 1 day (D) 1, in Part A and B of the study. All patients will receive lung SBRT on C1D15, C1D17, and C1D19 as per lung SBRT protocol (See Appendix 3). Although C1D1 can occur +/- 3 days, C1D15, C1D17, and C1D19, must be scheduled for a Monday, Wednesday and Friday, respectively. Patients in part A will receive lung SBRT dosed at 30 Gy in 3# in cohort 1, or 54 Gy in 3# in cohort 2. Patients in Part B will receive the RP2D of lung SBRT, determined in Part A. All patients in Part A and Part B will receive pembrolizumab dosed at 200 mg every 3 weeks, until disease progression, unacceptable toxicities, the patient withdraws consent from the trial, or the patient has completed 24 months of treatment.

In the dose escalation phase, a minimum of 3 patients will be required per dose level being assessed. A minimum gap of 1 week will be left between the treatment of the first and the second, and between the second and the third patients with the combination of pembrolizumab and lung SBRT to mitigate against multiple patients suffering from acute toxicity. The DLT period for this study is 12 weeks from the last dose of lung SBRT (i.e. at C6D1). The dose escalation will be considered by the Safety Review Committee (SRC) once the 3rd or 6th patient in the cohort has completed the DLT period. If no DLT is observed at a dose level, then lung SBRT will be dose escalated to the next dosing level (see Table 1). If 1 out of 3 patients experience a DLT, then the cohort will be expanded to 6 patients. If 1 in 6 patients experience a DLT, then the dose will be escalated to the next dosing level. However, if ≥ 2 in 6 patients experience a DLT then the maximum administered dose (MAD) will have been reached, and the RP2D will be the previous dosing level that will be used for the dose expansion cohorts. If the MAD is seen at dose level 1 then the study will be terminated. While waiting for 3 or 6 patients to complete the DLT period, no additional patients will be recruited. Further patients can only be recruited after the SRC has reviewed the toxicity data for the cohort and taken a decision to dose escalate to the next cohort or expand the current cohort to 6 patients.

Once the MTD has been determined the trial enters the dose expansion phase (unless the MTD is dose level 1). Here, 12 patients will be treated with the RP2D of SBRT combined with pembrolizumab.

If there is ongoing clinical benefit at 24 months, the CI/PI will need to discuss with the sponsor and MSD, on a case by case basis for the continuation of pembrolizumab.

ELIGIBILITY:
Inclusion Criteria:

1. Patients should be ≥18 years old on the day of signing the informed consent.
2. Patients must have a histological or cytological diagnosis of NSCLC.
3. Patients should have non-radically treatable stage IIIB or IV disease.
4. Patients must have measurable disease as assessed by RECIST v1.1.
5. Patients must have had disease progression or be intolerant of standard first line palliative chemotherapy for non-small cell lung cancer. If they are known to have a driver mutation for which there is a small molecule targeted therapy, they must have had disease progression or be intolerant of this.
6. Patient should have an ECOG performance status 0-1.
7. Patients should be able to tolerate a course of stereotactic radiotherapy as assessed by the investigator.
8. Patients should have disease within the lung, away from critical structures, suitable for treatment to part of a lesion with lung SBRT.
9. Patients must have adequate organ function including MRC dyspnoea score <3 and adequate baseline lung function tests, with an FEV1 > 0.8L or >30% of predicted and a TLCO > 30%
10. Demonstrate adequate organ function (based on bloods within 10 days of C1D1).
11. Have provided tissue from an archival tissue sample or newly obtained tissue sample.
12. Female patient of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication (C1D1). If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
13. Female patients of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication. Patients of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year.
14. Male patients should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy.
15. Be willing to provide informed consent for the trial.

Exclusion Criteria:

1. Patients who have taken any investigational medicinal product or have used an investigational device within 4 weeks of the first dose of pembrolizumab. Patients may participate in additional observational studies.
2. Patients who have received prior chemotherapy, targeted small molecule therapy or radiotherapy within 4 weeks prior to the first dose of pembrolizumab.
3. Patients with a diagnosis of immunodeficiency or be receiving systemic steroid therapy (>7.5 mg of prednisone / >1 mg of dexamethasone or their equivalent dose) or any other form of immunosuppressive therapy within 7 days prior to the first dose.
4. Patients with evidence of active autoimmune disease requiring systemic treatment within the past 3 months or a documented history of clinically severe autoimmune disease, or a syndrome that requires systemic steroids or immunosuppressive agents.
5. Patients who have received prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-Cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) antibody (including ipilimumab or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways).
6. Patients with evidence of active central nervous system (CNS) metastases and/or carcinomatous meningitis. Patients with previously treated brain metastases may participate provided the brain metastases are stable and there is no evidence of new or enlarging brain metastases.
7. Patients who have had previous radiotherapy to the lung or other neighbouring region that would preclude the safe administration of lung SBRT.
8. Patients with evidence of interstitial lung disease, or history of pneumonitis (including non-infectious pneumonitis) that required steroids, or current pneumonitis (including non-infectious pneumonitis).
9. Patients with evidence of additional malignancy that is progressing or requires active treatment.
10. Patients with a history or current evidence of any condition, therapy, or laboratory abnormality that might confound trial results, interfere with the patient's participation or is not in the best interest of the patient.
11. Patients with psychiatric or substance abuse disorders that would interfere with patient's participation.
12. Patients who are pregnant / breastfeeding or expecting to conceive within the duration of the trial, starting with the screening visit through 120 days after the last dose.
13. Patients with a history of HIV, HIV 1/2 antibodies, Hepatitis B or Hepatitis C.
14. Patients who have received a live vaccine within 30 days prior to the first dose of trial treatment.
15. Patients with known hypersensitivity to the active substance pembrolizumab or to any of the excipients listed in the SmPC.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-07-08 (Actual); Study Completion 2019-07-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fiona McDonald, MD, Study Chair — Royal Marsden NHS Foundation Trust
Locations (1):
- Royal Marsden NHS Foundation Trust, Sutton, Surrey, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: During the period between June 2018 and January 2019, 2 patients were recruited to the study at the Royal Marsden Hospital in the United Kingdom.
Groups:
- Dose Escalation Cohort - DOSE LEVEL 1: Intervention: One dose pembrolizumab 200 mg (week 1) followed by lung Stereotactic Body Radiotherapy (SBRT) 30 Gy 3 fractions (#) in week 3. Treatment with pembrolizumab 200 mg will be continued given every 3 weeks.
  Stereotactic Body Radiotherapy (SBRT) 30 Gy 3 fractions (#): Stereotactic Body Radiotherapy (SBRT) dosed at 30 Gy in 3 fractions (#) in week 3
  Pembrolizumab: Pembrolizumab in week 1 dosed at 200 mg (prior to SBRT) and then treatment with pembrolizumab will be continued dosed at 200 mg given every 3 weeks.
  Pembrolizumab administered as a 30-minute IV infusion.
- Dose Escalation Cohort - DOSE LEVEL 2: Intervention: One dose of pembrolizumab 200 mg (week 1) followed by lung Stereotactic Body Radiotherapy (SBRT) 54 Gy 3 fractions (#) in week 3. Treatment with pembrolizumab 200 mg will be continued given every 3 weeks.
  Stereotactic Body Radiotherapy (SBRT) 54 Gy 3 fractions (#): Stereotactic Body Radiotherapy (SBRT) dosed at 54 Gy in 3 fractions (#) in week 3
  Pembrolizumab: Pembrolizumab in week 1 dosed at 200 mg (prior to SBRT) and then treatment with pembrolizumab will be continued dosed at 200 mg given every 3 weeks.
  Pembrolizumab administered as a 30-minute IV infusion.
- Part B - Expansion Cohort: Intervention: One dose of pembrolizumab 200 mg (week 1) followed in by lung Stereotactic Body Radiotherapy (SBRT) dosed at the maximum tolerated dose determined in Part A in week 3, dosed at the maximum tolerated dose determined in Part A. Treatment with pembrolizumab 200 mg will be continued given every 3 weeks.
  Stereotactic Body Radiotherapy (SBRT) dosed at the maximum tolerated dose: Stereotactic Body Radiotherapy (SBRT) dosed at the maximum tolerated dose (MTD) determined in Part A in week 3
  Pembrolizumab: Pembrolizumab in week 1 dosed at 200 mg (prior to SBRT) and then treatment with pembrolizumab will be continued dosed at 200 mg given every 3 weeks.
  Pembrolizumab administered as a 30-minute IV infusion.
Period: Overall Study
Arm/Group | Dose Escalation Cohort - DOSE LEVEL 1 | Dose Escalation Cohort - DOSE LEVEL 2 | Part B - Expansion Cohort
Started | 2 | 0 | 0
Completed | 0 | 0 | 0
Not Completed | 2 | 0 | 0
Not completed — Lack of Efficacy | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Population: No participants were recruited to Dose Level 2 of Dose Escalation Cohort and to Expansion Cohort.
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose Escalation Cohort - DOSE LEVEL 1 | Dose Escalation Cohort - DOSE LEVEL 2 | Part B - Expansion Cohort | Total
Number analyzed (Participants) | 2 | 0 | 0 | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 |  |  | 0
  Between 18 and 65 years | 0 |  |  | 0
  >=65 years | 2 |  |  | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 |  |  | 1
  Male | 1 |  |  | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  |  | 0
  Asian | 0 |  |  | 0
  Native Hawaiian or Other Pacific Islander | 0 |  |  | 0
  Black or African American | 0 |  |  | 0
  White | 2 |  |  | 2
  More than one race | 0 |  |  | 0
  Unknown or Not Reported | 0 |  |  | 0
Region of Enrollment [Number; unit: participants]
  United Kingdom | 2 |  |  | 2
Eastern Cooperative Oncology Group (ECOG) [Count of Participants; unit: Participants]
  0 = Normal activity. | 0 |  |  | 0
  1 = Symptoms but ambulatory. | 2 |  |  | 2

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients With Dose Limiting Toxicity
Description: Proportion of all treated patients who have experience at least one Dose Limiting Toxicity (DLT). DLT is assessed using NCI CTCAE v4.0 and defined as any one or more of: neutropenia with fever grade >=3; thrombocytopenia with bleeding grade >=3; any grade >=3 non-haematological toxicity which is definitely, probably, or possibly related to the trial treatment.
Time Frame: From first dose of Pembrolizumab to 12 weeks from the last dose of lung SBRT
Population: All patients who completed the DLT period
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Escalation Cohort - DOSE LEVEL 1 | Dose Escalation Cohort - DOSE LEVEL 2 | Part B - Expansion Cohort
Number analyzed (Participants) | 2 | 0 | 0
Participants | 0 |  |

2. Secondary Outcome: Acute Toxicity Rate
Description: Percentage of patients any acute toxicity, by worst grade as assessed using CTCAE v4.0
Time Frame: From first dose of Pembrolizumab to 12 weeks from the last dose of lung SBRT
Population: All patients who recieved at least one dose of trial treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Escalation Cohort - DOSE LEVEL 1 | Dose Escalation Cohort - DOSE LEVEL 2 | Part B - Expansion Cohort
Number analyzed (Participants) | 2 | 0 | 0
Participants
  Patients with max grade 3 toxicity | 0 |  |
  Patients with max grade 2 toxicity | 1 |  |
  Patients with max grade 1 toxicity | 1 |  |

3. Secondary Outcome: Late Toxicity Rate
Description: Percentage of patients with any late toxicity, by worst grade as assessed using CTCAE v4.0
Time Frame: Assessed at start of each 21 day pembrolizumab cycle, starts from 12 weeks after last fraction of lung SBRT and ends 28 days after last on-trial dose of pembrolizumab (treatment ended at disease progression for all trial patients), up to 6 months
Population: All patients who received at least one dose of pembrolizumab and one fraction of radiotherapy
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Escalation Cohort - DOSE LEVEL 1 | Dose Escalation Cohort - DOSE LEVEL 2 | Part B - Expansion Cohort
Number analyzed (Participants) | 2 | 0 | 0
Participants
  Patients with max grade 3 toxicity | 1 |  |
  patients with max grade 2 toxicity | 0 |  |
  Patients with max grade 1 toxicity | 1 |  |

4. Secondary Outcome: Overall Response Rate
Description: Count of patients with best overall response of complete or partial response at any time, assessed using RECIST v1.1
Time Frame: Response assessed from start of pembrolizumab, every 9 weeks for the first 6 months, then every 12 weeks thereafter, until the first instance of documented disease progression (occurred no later than 7 months from start of treatment for all patients)
Population: All patients with at least one dose of trial treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Escalation Cohort - DOSE LEVEL 1 | Dose Escalation Cohort - DOSE LEVEL 2 | Part B - Expansion Cohort
Number analyzed (Participants) | 2 | 0 | 0
Participants | 0 |  |

5. Secondary Outcome: Disease Control Rate
Description: Count of patients with best overall response at any time of complete or partial response, or stable disease, assessed by RECIST v1.1
Time Frame: as for outcome 4
Population: All patients with at least one dose of trial treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Escalation Cohort - DOSE LEVEL 1 | Dose Escalation Cohort - DOSE LEVEL 2 | Part B - Expansion Cohort
Number analyzed (Participants) | 2 | 0 | 0
Participants | 2 |  |

6. Secondary Outcome: Overall Response Rate (irRECIST)
Description: Count of patients with best response of complete or partial response, assessed using Immune Related Response Criteria (irRC) as defined by: Wolchok JD et al. Guidelines for the evaluation of immune therapy activity in solid tumors: Immune related response criteria. Clin Cancer Res 2009;15(23):7412. (72)
Time Frame: Response assessed from start of pembrolizumab, every 9 weeks for the first 6 months, then every 12 weeks thereafter, until the first instance of documented disease progression, start of new anti-cancer treatment, death or end of study
Population: No patients were assessed using irRECIST, as the study was terminated early after treating a total of two patients. Although imaging was performed and standard response measurement were done as per RECIST, the sum of the products of the two longest perpendicular diameters as required by irRECIST was not measured.
Arm/Group | Dose Escalation Cohort - DOSE LEVEL 1 | Dose Escalation Cohort - DOSE LEVEL 2 | Part B - Expansion Cohort
Number analyzed (Participants) | 0 | 0 | 0

7. Secondary Outcome: Frequency of PD-1/PD-L1 Expression
Description: PD-1/PD-L1 expression distribution in responders and non-responders
Time Frame: Response to be defined as per previous endpoint, PD1/PD-L1 to be measured at study entry
Population: The planned tissue evaluation for PD1/PD-L1 status was not done (and will not be performed in future) as the study was terminated early after treating a total of two patients
Arm/Group | Dose Escalation Cohort - DOSE LEVEL 1 | Dose Escalation Cohort - DOSE LEVEL 2 | Part B - Expansion Cohort
Number analyzed (Participants) | 0 | 0 | 0

8. Secondary Outcome: Overall Survival at Six Months
Description: Count of patients known to be alive at six months
Time Frame: 6 months after last dose of lung SBRT
Population: All patients assessed for survival at six months following last dose of lung SBRT
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Escalation Cohort - DOSE LEVEL 1 | Dose Escalation Cohort - DOSE LEVEL 2 | Part B - Expansion Cohort
Number analyzed (Participants) | 2 | 0 | 0
Participants | 2 |  |

9. Secondary Outcome: Overall Survival at 12 Months
Description: Count of patients known to be alive at 12 months
Time Frame: 12 months after last dose of lung SBRT
Population: All patients assessed for survival at 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Escalation Cohort - DOSE LEVEL 1 | Dose Escalation Cohort - DOSE LEVEL 2 | Part B - Expansion Cohort
Number analyzed (Participants) | 1 | 0 | 0
Participants | 1 |  |

10. Secondary Outcome: Progression Free Survival at 6 Months
Description: Count of patients known to be alive and free from progression at 6 months
Time Frame: 6 months after last dose of lung SBRT
Population: All patients assessed for progression and survival at 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Escalation Cohort - DOSE LEVEL 1 | Dose Escalation Cohort - DOSE LEVEL 2 | Part B - Expansion Cohort
Number analyzed (Participants) | 2 | 0 | 0
Participants | 1 |  |

11. Secondary Outcome: Progression Free Survival at 12 Months
Description: Count of patients known to be alive and free from progression at 12 months
Time Frame: 12 months after last dose of lung SBRT
Population: All patients assessed for progression and survival at 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Escalation Cohort - DOSE LEVEL 1 | Dose Escalation Cohort - DOSE LEVEL 2 | Part B - Expansion Cohort
Number analyzed (Participants) | 2 | 0 | 0
Participants | 0 |  |

ADVERSE EVENTS:
Time Frame: Adverse events were recorded from confirmation of entry into the trial at the start of each 21 day pembrolizumab cycle, until the patients 30 day safety follow up visit. All cause mortality was recorded up to 12 months after last dose of lung SBRT.
Description: No patients were recruited to Dose Level 2 of Dose Escalation Cohort and to Expansion Cohort, therefore number of patients at risk is 0 for these.
Arm/Group | Dose Escalation Cohort - DOSE LEVEL 1 | Dose Escalation Cohort - DOSE LEVEL 2 | Part B - Expansion Cohort
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 2/2 | 0/0 | 0/0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Escalation Cohort - DOSE LEVEL 1 (N=2) | Dose Escalation Cohort - DOSE LEVEL 2 (N=0) | Part B - Expansion Cohort (N=0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | NA | NA
Dyspepsia (Gastrointestinal disorders) | 1 (1) | NA | NA
Abdominal pain (Gastrointestinal disorders) | 1 (1) | NA | NA
Nausea (Gastrointestinal disorders) | 1 (1) | NA | NA
Fatigue (General disorders) | 2 (2) | NA | NA
Flu like symptoms (General disorders) | 1 (1) | NA | NA
Urinary tract infection (Infections and infestations) | 1 (1) | NA | NA
Upper respiratory infection (Infections and infestations) | 1 (1) | NA | NA
Bruising (Injury, poisoning and procedural complications) | 1 (1) | NA | NA
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | NA | NA
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | NA | NA
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | NA | NA
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 (2) | NA | NA
Headache (Nervous system disorders) | 1 (1) | NA | NA
Dysgeusia (Nervous system disorders) | 1 (1) | NA | NA
Dizziness (Nervous system disorders) | 1 (1) | NA | NA
Acute kidney injury (Renal and urinary disorders) | 1 (1) | NA | NA
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | NA | NA
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | NA | NA
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | NA | NA
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | NA | NA
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 1 (1) | NA | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-14): https://cdn.clinicaltrials.gov/large-docs/56/NCT03436056/Prot_SAP_000.pdf